CLINICAL TRIAL: NCT03535857
Title: Effectiveness of Bilateral PTNS Compared to Unilateral PTNS for the Treatment of Overactive Bladder/Urge Incontinence
Acronym: BUTTON
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Challenges with recruitment
Sponsor: Gnankang Sarah Napoe (Other)
Responsible Party: Sponsor-Investigator, Gnankang Sarah Napoe, Assistant Professor, University of Pittsburgh
Organization: University of Pittsburgh (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: STUDY19100230
Record Dates: First submitted 2018-05-08; First posted 2018-05-24 (Actual); Results first posted 2025-04-06 (Actual); Last update posted 2025-04-15 (Actual); Status verified 2025-04

CONDITIONS: Overactive Bladder Syndrome; Urinary Incontinence, Urge
Keywords: overactive bladder; OAB; urge urinary incontinence; PTNS
MeSH Terms: conditions — Urinary Incontinence, Urge; Urinary Bladder, Overactive

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- Unilateral PTNS (Active Comparator): 34 gauge needle inserted 3cm above the medial ankle on the ankle, and cables are connected to the PTNS stimulator device. Stimulation is provided, per manufacturer directions, over a 30-minute treatment period
  Interventions: Device: PTNS
- Bilateral PTNS (Experimental): 34 gauge needle inserted 3cm above the medial ankle on both ankles, and cables are connected to the PTNS stimulator device. Stimulation is provided, per manufacturer directions, over a 30-minute treatment period
  Interventions: Device: PTNS

INTERVENTIONS:
Device: PTNS — Use of PTNS on the ankle for 30 minutes

SUMMARY:
This study is designed to evaluate whether bilateral Posterior Tibial Nerve Stimulation is more effective than unilateral Posterior Tibial Nerve Stimulation at treating overactive bladder and urge urinary incontinence

DETAILED DESCRIPTION:
Percutaneous tibial nerve stimulation (PTNS) is an accepted treatment for overactive bladder that can be accomplished in the office with minimal side effects. It is currently carried out by stimulating one of the posterior tibial nerves unilaterally. The aim of this study is to determine whether bilateral percutaneous tibial nerve stimulation is more effective than unilateral stimulation. Patients with a diagnosis of overactive bladder who have previously failed lifestyle changes and/or pharmacologic therapy will be offered percutaneous tibial nerve stimulation. Enrolled patients will be randomized into two groups. The control group will receive the traditional unilateral treatment of PTNS. The intervention group will receive bilateral PTNS treatment. Intervention success will be measured by improvement in overactive bladder symptoms assessed by improvement in the scores on the overactive bladder questionnaire symptoms bother and decrease in number of voids, nocturia episodes and incontinence episodes as reported in the voiding diary

ELIGIBILITY:
Inclusion Criteria:

1. Female patients over the age of 18 who have previously tried and failed, or were unable to tolerate, behavioral therapy
2. Patients who consent to participate in the study
3. Patients on pharmacologic therapy at the time of recruitment can continue their treatment

Exclusion Criteria:

1. Pregnant patients
2. Patients with pacemakers of implantable defibrillators
3. Patients with neurogenic bladder
4. Patients who have received Botox or have an implant for sacral nerve stimulation
5. Patients with uncontrolled bleeding disorder
6. Patients with unhealed ulcers or with leg edema surrounding medial malleolus

Ages: 18 Years to 99 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2018-04-17 (Actual); Primary Completion 2023-09-08 (Actual); Study Completion 2023-09-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: G. Sarah Napoe, MD, Principal Investigator — University of Pittsburgh; Kyle Wohlrab, MD, Principal Investigator — Women and Infants Hospital of Rhode Island
Locations (2):
- United States (2):
  - Gnankang Sarah Napoe, Pittsburgh, Pennsylvania
  - WIHRI, Providence, Rhode Island

IPD SHARING:
Plan to Share IPD: No
No plan to share IPD

REFERENCES:
- [Derived] Napoe GS, Hall E, Dasgupta P, Myers DL, Wohlrab KJ. Randomized trial of unilateral versus bilateral percutaneous tibial nerve stimulation for the treatment of overactive bladder. World J Urol. 2025 Dec 4;44(1):15. doi: 10.1007/s00345-025-06107-0. PMID 41342952

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Unilateral PTNS | Bilateral PTNS
Started | 18 | 18
Completed | 13 | 16
Not Completed | 5 | 2

BASELINE CHARACTERISTICS:
Groups:
- Bilateral PTNS: PTNS: Use of PTNS on both ankles for 30 minutes
- Total: Total of all reporting groups
Arm/Group | Unilateral PTNS | Bilateral PTNS | Total
Number analyzed (Participants) | 18 | 18 | 36
Age, Customized [Mean (Standard Deviation); unit: years]
  Age | 68.1 (13.8) | 69.4 (11.4) | 68.7 (12.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 18 | 18 | 36
  Male | 0 | 0 | 0
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
On Overactive bladder (OAB) Medications [Number; unit: participants] | 6 | 4 | 10
History of Diabetes mellitus [Number; unit: participants] | 2 | 7 | 9
Overactive bladder questionnaire short form (OABq SF) Score [Mean (Standard Deviation); unit: units on a scale] — Population: Missing data
  units on a scale
    number analyzed (Participants) | 17 | 18 | 35
    (all) | 64.6 (21.6) | 56.1 (26.2) | 60.4 (24.1)
Incontinence Impact Questionnaire (IIQ) Score [Mean (Standard Deviation); unit: units on a scale] — Population: Missing data
  units on a scale
    number analyzed (Participants) | 17 | 18 | 35
    (all) | 49.5 (29.7) | 59.8 (23.6) | 54.8 (26.9)
Daily Incontinence Episodes [Mean (Standard Deviation); unit: Incontinence episodes] — Population: Missing data
  Incontinence episodes
    number analyzed (Participants) | 16 | 17 | 33
    (all) | 2.3 (2.4) | 2.6 (2.0) | 2.5 (2.2)
Nocturia Episodes [Mean (Standard Deviation); unit: Nocturia episodes] — Population: Missing data
  Nocturia episodes
    number analyzed (Participants) | 8 | 9 | 17
    (all) | 1.7 (1.4) | 1.7 (1.9) | 1.7 (1.6)
Daily voids [Mean (Standard Deviation); unit: Daily voids] — Population: Missing data
  Daily voids
    number analyzed (Participants) | 16 | 17 | 33
    (all) | 9.8 (3.2) | 9.6 (4.1) | 9.7 (3.7)

OUTCOME MEASURES:

1. Primary Outcome: Change in Overactive Bladder Questionnaire Score From Baseline to 12 Weeks or Last Measurement
Description: Overactive Bladder questionnaire short form (OABqSF) symptom severity questionnaire was administered at baseline, 4 weeks, 8 weeks then 12 weeks. The OABqSF score ranges from 0 to 100. Those with more bothersome symptoms have higher scores.
  The investigators expected more improvement in symptoms from participants receiving bilateral stimulation compared to those with unilateral stimulation.
Time Frame: 12 weeks or last measurement
Population: Analysis was performed on all enrolled participants data available even if the participant withdrew from study prior to completion of study.
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Unilateral PTNS Change in Overactive Bladder Questionnaire Short Form Score: Change in overactive bladder symptom severity was measured by comparing last overactive bladder questionnaire score to overactive bladder questionnaire score at baseline for one ankle stimulation
- Bilateral PTNS Change in Overactive Bladder Questionnaire Short Form Score: Change in overactive bladder symptom severity was measured by comparing last overactive bladder questionnaire score to overactive bladder questionnaire score at baseline for two ankle stimulation
Arm/Group | Unilateral PTNS Change in Overactive Bladder Questionnaire Short Form Score | Bilateral PTNS Change in Overactive Bladder Questionnaire Short Form Score
Number analyzed (Participants) | 17 | 17
score on a scale | -17.8 (24.7) | -23.5 (29.3)
Statistical Analysis 1: Comparison: Unilateral PTNS Change in Overactive Bladder Questionnaire Short Form Score vs Bilateral PTNS Change in Overactive Bladder Questionnaire Short Form Score; Test type: Superiority; p = 0.546, Pairwise t- test; Mean Difference (Final Values) = 5.7

2. Secondary Outcome: Change in Daily Number of Voids From Baseline to 12 Weeks or Last Measurement
Description: The change in number of voids was obtained by comparing number of voids at 12 weeks or last measurement compared to baseline number of voids.
Time Frame: 12 weeks or last measurement
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Number of daytime voids
Groups:
- Unilateral PTNS Change in Number of Daily Voids: Change in number of voids defined as number of voids at completion of PTNS (12 weeks or last measurement) compared to baseline number of voids for unilateral stimulation
- Bilateral PTNS Change in Number of Daily Voids: Change in number of voids defined as number of voids at completion of PTNS (12 weeks or last measurement) compared to baseline number of voids for bilateral stimulation
Arm/Group | Unilateral PTNS Change in Number of Daily Voids | Bilateral PTNS Change in Number of Daily Voids
Number analyzed (Participants) | 16 | 17
Number of daytime voids | -0.2 (3.3) | -1.3 (2.6)

3. Secondary Outcome: Change in Number of Incontinence Episodes Per 24 Hours From Baseline to 12 Weeks or Last Measurement
Description: Change in number of incontinence episodes defined as number of incontinence episodes at completion of PTNS (12 weeks or last measurement) compared to baseline number of incontinence episodes.
Time Frame: 12 weeks or last measurement
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Number of incontinence episodes
Groups:
- Unilateral PTNS Change in Number of Incontinence Episodes: Change in number of incontinence episodes defined as number of incontinence episodes at completion of PTNS (12 weeks or last measurement) compared to baseline number of incontinence episodes for one ankle stimulation
- Bilateral PTNS Change in Number of Incontinence Episodes Per 24 Hours: Change in number of incontinence episodes defined as number of incontinence episodes at completion of PTNS (12 weeks or last measurement) compared to baseline number of incontinence episodes for two ankle stimulation
Arm/Group | Unilateral PTNS Change in Number of Incontinence Episodes | Bilateral PTNS Change in Number of Incontinence Episodes Per 24 Hours
Number analyzed (Participants) | 16 | 17
Number of incontinence episodes | -0.3 (3.6) | -1.2 (1.3)

4. Secondary Outcome: Change in Nocturia Episodes From Baseline to 12 Weeks or Last Measurement
Description: Change in number of nocturia episodes defined as number of nighttime voids at completion of PTNS (12 weeks or last measurement) compared to baseline number of nighttime voids.
Time Frame: 12 weeks or last measurement
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Number of nighttime voids
Groups:
- Unilateral PTNS Nocturia Episodes at Last Measurement: Change in number of nocturia episodes defined as number of nighttime voids at completion of PTNS (12 weeks or last measurement) compared to baseline number of nighttime voids for one ankle stimulation
- Bilateral PTNS Nocturia Episodes at Last Measurement: Change in number of nocturia episodes defined as number of nighttime voids at completion of PTNS (12 weeks or last measurement) compared to baseline number of nighttime voids for two ankle stimulation
Arm/Group | Unilateral PTNS Nocturia Episodes at Last Measurement | Bilateral PTNS Nocturia Episodes at Last Measurement
Number analyzed (Participants) | 10 | 9
Number of nighttime voids | -0.1 (1.1) | -0.8 (1.4)

5. Secondary Outcome: Impact of Treatment on Quality of Life From Baseline to 12 Weeks or Last Measurement
Description: The incontinence impact questionnaire was used to measure the impact on quality of life. The questionnaire score ranges from 0 to 100 with higher scores indicating worse quality of life.
Time Frame: 12 weeks or last measurement
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Unilateral PTNS Incontinence Impact Questionnaire-7 Score Change: Impact of treatment on quality of life was measured by comparing the last incontinence impact questionnaire score to the baseline incontinence impact questionnaire score for one ankle stimulation
- Bilateral PTNS Incontinence Impact Questionnaire-7 Score Change: Impact of treatment on quality of life was measured by comparing the last incontinence impact questionnaire score to the baseline incontinence impact questionnaire score for two ankle stimulation
Arm/Group | Unilateral PTNS Incontinence Impact Questionnaire-7 Score Change | Bilateral PTNS Incontinence Impact Questionnaire-7 Score Change
Number analyzed (Participants) | 16 | 17
score on a scale | -12.8 (24.7) | -19.3 (18.9)

ADVERSE EVENTS:
Time Frame: 12 weeks
Groups:
- Unilateral PTNS: One ankle stimulation
- Bilateral PTNS: Two ankle stimulation
Arm/Group | Unilateral PTNS | Bilateral PTNS
All-Cause Mortality (participants affected / at risk) | 0/18 | 0/18
Serious Adverse Events (participants affected / at risk) | 0/18 | 0/18
Other Adverse Events (participants affected / at risk) | 0/18 | 0/18

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2024-04-30): https://cdn.clinicaltrials.gov/large-docs/57/NCT03535857/Prot_SAP_001.pdf